CLINICAL TRIAL: NCT01616277
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-06252616 In Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate The Safety And Tolerability Of PF-06252616 In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B5161001
Record Dates: First submitted 2012-05-25; First posted 2012-06-11 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — domagrozumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Placebo Comparator)
  Interventions: Biological: PF-06252616; Drug: Placebo
- 2 (Placebo Comparator)
  Interventions: Biological: PF-06252616; Drug: Placebo
- 3 (Placebo Comparator)
  Interventions: Biological: PF-06252161; Drug: Placebo
- 4 (Placebo Comparator)
  Interventions: Biological: PF-06252616; Drug: Placebo
- 5 (Placebo Comparator): Repeat dose of PF-06252616, IV infusion, single dose - 10.0 miligram per kilogram
  Interventions: Biological: PF-06252616; Drug: Placebo
- 6 (Placebo Comparator)
  Interventions: Biological: PF-06252616; Drug: Placebo
- 7 (Placebo Comparator)
  Interventions: Biological: PF-06252616; Drug: Placebo

INTERVENTIONS:
Biological: PF-06252616 — 1.0 milligram per kilogram of PF-06252616, IV infusion, single dose
  Arms: 1
Drug: Placebo — Placebo for PF-06252616, IV infusion, single dose
  Arms: 1
Biological: PF-06252616 — 3.0 milligram per kilogram of PF-06252616, IV infusion, single dose
  Arms: 2
Drug: Placebo — Placebo for PF-06252616, IV infusion, single dose
  Arms: 2
Biological: PF-06252161 — 10.0 milligram per kilogram of PF-06252616, IV infusion, single dose
  Arms: 3
Drug: Placebo — Placebo for PF-06252616, IV infusion, single dose
  Arms: 3
Biological: PF-06252616 — 3.0 milligram per kilogram of PF-06252616, Subcutaneous injection, single dose
  Arms: 4
Drug: Placebo — Placebo for PF-06252616, Subcutaneous injection, single dose
  Arms: 4
Biological: PF-06252616 — 10.0 miligram per kilogram of PF-06252616, IV infusion, repeat dose
  Arms: 5
Drug: Placebo — Placebo for PF-06252616, IV infusion, repeat dose
  Arms: 5
Biological: PF-06252616 — 20.0 milligram per kilogram of PF-06252616, IV infusion, single dose
  Arms: 6
Drug: Placebo — Placebo for PF-06252616, IV infusion, single dose
  Arms: 6
Biological: PF-06252616 — 40.0 milligram per kilogram of PF-06252616, IV infusion, single dose
  Arms: 7
Drug: Placebo — Placebo for PF-06252616, IV infusion, single dose
  Arms: 7

SUMMARY:
The purpose of this study is to determine if the study drug, PF-06252616 is safe and well tolerated when given to adult healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Single Dose Cohorts-Healthy male and/or female non-child bearing subjects between the ages of 18 and 55 years, inclusive.
* Repeat Dose Cohort-Healthy male and/or female non-child bearing subjects between the ages of 18 and less than 65 years, inclusive.

Exclusion Criteria:

* Presence or history of muscle disease (eg, polymyositis or rhabdomyolysis).
* Weight loss or gain of >5% within 30 days of Screening, as reported by subject.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, immunologic, metabolic urologic, dermatologic, renal, allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) and any other major disease.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related Adverse Events. | Day 197
Severity of treatment related Adverse Events. | Day 197
Incidence of abnormal lab findings. | Day 197
Magnitude of abnormal lab findings. | Day 197
Abnormal and clinically relevant changes in Blood Pressure. | Day 197
Abnormal and clinically relevant changes in Pulse Rate. | Day 197
Abnormal and clinically relevant changes in Respiratory Rate. | Day 197
Abnormal and clinically relevant changes in temperature. | Day 197
Abnormal and clinically relevant changes in ECG parameters. | Day 197

SECONDARY OUTCOMES:
PF-06252616 concentration in serum as measured by a validated PK assay for Cmax (maximum concentration) | Through Day 197 post dosing
Pharmacodynamic activity as measured by serum concentrations of GDF-8 (myostatin) as measured by a GDF-8 assay | Through Day 197 post dosing
Incidence of development of anti-drug antibody (ADA) as measured by an ADA assay | Through Day 197 post dosing
Pharmacologic activity as measured by the percent change in lean body mass as measured by DXA | Through Day 113 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for Tmax (time to reach maximum concentration) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for AUCinf (area under the curve serum concentration-time profile from time zero to infinity | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for AUClast (area under the curve serum concentration from time zero to the time of the last quantifiable concentration) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for t1/2 (half-life time for the serum concentration to decrease by half). | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for AUCτ (area under the curve serum concentration by dose interval) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for MRT (mean residence time) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for CL (rate of clearance from serum) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for CLss (rate of steady state clearance from serum in the repeat dose cohort) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for Vz /F(volume of distribution is the theoretical volume which the total amount of drug would need to be uniformly distributed to produce the desired concentration of a drug.) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for Vss(volume of distribution is the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired concentration of a drug. | Through Day 197 post dosing
Steady state volume of distribution is the apparent volume of distribution at steady-state.) | Through Day 197 post dosing
PF-06252616 concentration in serum as measured by a validated PK assay for RAC (accumulation ratio for AUC) | Through Day 197 post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Wojciechowski J, Purohit VS, Harnisch LO, Dua P, Tan B, Nicholas T. Population PK and PD Analysis of Domagrozumab in Pediatric Patients with Duchenne Muscular Dystrophy. Clin Pharmacol Ther. 2022 Dec;112(6):1291-1302. doi: 10.1002/cpt.2747. Epub 2022 Oct 4. PMID 36104012
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5161001&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Safety%20And%20Tolerability%20Of%20PF-06252616%20In%20Healthy%20Subjects